CLINICAL TRIAL: NCT06643884
Title: A Phase 2, Open-Label, Dose Escalation Trial Assessing the Safety, Tolerability, and Treatment Effect of Belzupacap Sarotalocan (AU-011) With Suprachoroidal Administration in Subjects With Metastases to the Choroid
Brief Title: Suprachoroidal Administration in Subjects With Metastases to the Choroid
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aura Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AU-011-203
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Eye Cancer; Primary Cancer
Keywords: Choroidal Metastasis; Metastases to the Choroid; ocular; eye
MeSH Terms: conditions — Eye Neoplasms; Neoplasms | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (7):
- 80 micrograms of bel-sar (Experimental): 1 Cycle AU-011 with a dose of 80 micrograms
  Interventions: Drug: AU-011; Device: SCS Microinjector; Device: Laser
- 140 micrograms of bel-sar (Experimental): 1 Cycle AU-011 with a dose of 140 micrograms
  Interventions: Drug: AU-011; Device: SCS Microinjector; Device: Laser
- 200 micrograms of bel-sar with one cycle (Experimental): 1 Cycle AU-011 with a dose of 200 micrograms
  Interventions: Drug: AU-011; Device: SCS Microinjector; Device: Laser
- 200 micrograms of bel-sar with two cycles (Experimental): 2 Cycles AU-011 with a dose of 200 micrograms
  Interventions: Drug: AU-011; Device: SCS Microinjector; Device: Laser
- Observational (No Intervention): Subjects that meet trial inclusion, but do not meet criteria for enrollment into the bel-sar treatment cohorts, may be enrolled in this cohort. The observational cohort will not receive bel-sar treatment.
- 40 micrograms of bel-sar with one cycle (Experimental): 1 Cycle AU-011 with a dose of 40 micrograms
  Interventions: Drug: AU-011; Device: SCS Microinjector; Device: Laser
- 40 micrograms of bel-sar with two cycles (Experimental): 2 Cycles AU-011 with a dose of 40 micrograms
  Interventions: Drug: AU-011; Device: SCS Microinjector; Device: Laser

INTERVENTIONS:
Drug: AU-011 — AU-011 Via Suprachoroidal Administration with laser treatment
  Arms: 140 micrograms of bel-sar; 200 micrograms of bel-sar with one cycle; 200 micrograms of bel-sar with two cycles; 40 micrograms of bel-sar with one cycle; 40 micrograms of bel-sar with two cycles; 80 micrograms of bel-sar
Device: SCS Microinjector — Suprachoroidal Injection Device
  Arms: 140 micrograms of bel-sar; 200 micrograms of bel-sar with one cycle; 200 micrograms of bel-sar with two cycles; 40 micrograms of bel-sar with one cycle; 40 micrograms of bel-sar with two cycles; 80 micrograms of bel-sar
Device: Laser — Laser Administration
  Arms: 140 micrograms of bel-sar; 200 micrograms of bel-sar with one cycle; 200 micrograms of bel-sar with two cycles; 40 micrograms of bel-sar with one cycle; 40 micrograms of bel-sar with two cycles; 80 micrograms of bel-sar

SUMMARY:
The primary objective is to assess the safety and tolerability of bel-sar treatment in subjects with metastases to the choroid from any primary carcinoma.

DETAILED DESCRIPTION:
This is an open-label, dose escalation trial designed to assess safety and tolerability of 4 dose strengths and 1-2 cycles of bel-sar treatment in subjects with metastases to the choroid from any primary carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of Metastases to the Choroid, from a histopathologically or cytologically confirmed tumor.
* Have at least one Metastases to the Choroid in the study eye

Exclusion Criteria:

* Active ocular infection or disease.
* Must not have evidence of a primary tumor or metastatic lesion in the brain requiring treatment with radiation therapy per the primary treating oncologist's assessment.
* Must not be planning or expecting to switch/add systemic antineoplastic therapies during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in choroidal tumor thickness on B-scan ultrasonography (B-scan) 4 weeks after completion of treatment. | 4 weeks after completion of treatment
  B-Scan Ultrasonography
Change from baseline in choroidal tumor largest basal diameter (LBD) on fundus photos 4 weeks after completion of treatment. | 4 weeks after completion of treatment
  Fundus photos

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Aura Biosciences
Locations (10):
- United States (10):
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Kellogg Eye Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cole Eye Institute, Cleveland, Ohio
  - Shields and Shields, PC, Philadelphia, Pennsylvania
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Consultants of Texas, Bellaire, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No